CLINICAL TRIAL: NCT01768858
Title: Assessment of Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, Plaque Psoriasis, Crohn's Disease and Ulcerative Colitis Patients´ Adherence Attitudes to Maintenance Therapy With a Scheduled Adalimumab Treatment in Routine Clinical Practice
Acronym: Adherence
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: Raffeiner GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-562
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Crohn´s Disease; Ulcerative Colitis; Plaque Psoriasis
Keywords: Arthritis; Morbus Crohn; Adherence; Spondylitis; Ulcerative colitis; Monoclonals; Rheumatoid; Antibodies; Ankylosing; Plaque psoriasis; Psoriatic; Crohn´s disease; Antirheumatic Agents
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Crohn Disease; Colitis, Ulcerative; Arthritis; Spondylitis | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants receiving adalimumab: Adults with rheumatoid arthritis (RA), psoriatic arthritis (PsA), ankylosing spondylitis (AS), plaque psoriasis (PS), Crohn´s disease (CD), or ulcerative colitis (UC) received 40 mg adalimumab every two weeks.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab administered by subcutaneous injection, via pre-filled syringe or autoinjector pen
  Other Names: Humira; ABT-D2E7

SUMMARY:
The purpose of this non-interventional, multicenter, post-marketing observational study (PMOS) was to assess rheumatoid arthritis (RA), psoriatic arthritis (PsA), ankylosing spondylitis (AS), plaque psoriasis (PS), Crohn's disease (CD) and ulcerative colitis (UC) patients' adherence attitudes (beliefs) to maintenance therapy with adalimumab monotherapy or combination therapy with methotrexate (in participants with RA) and to investigate whether there were correlations between such beliefs and adherence to maintenance treatment.

DETAILED DESCRIPTION:
Adalimumab was prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication. The assignment of a participant to an adalimumab-containing regimen was decided in advance and was to be current practice. The prescribing of adalimumab was clearly separated from the decision to include the participant in the study. Participants were observed for a maximum of 12 months, with a total of 5 study visits (Screening = Visit 1).

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age with rheumatoid arthritis (RA), psoriatic arthritis (PsA), ankylosing spondylitis (AS), plaque psoriasis (PS), Crohn´s disease (CD), or ulcerative colitis (UC)
* Participants must fulfill international and national guidelines for the use of a biologic disease-modifying antirheumatic drug (bDMARD) in RA, PsA, AS, PS, CD, or UC (chest X-ray and interferon gamma release assay (IGRA) or purified protein derivative (PPD) skin test negative for tuberculosis)
* In addition one of the following criteria must be fulfilled:

  1. unsatisfactory DMARD response defined as treatment failure with at least two DMARDs including methotrexate in participants with RA or PsA
  2. unsatisfactory nonsteroidal anti-inflammatory drug (NSAID) response in participants with AS
  3. unsatisfactory response to prior bDMARDs in participants with RA, PsA, or AS
  4. unsatisfactory response to, contraindication to, or intolerance to other systemic therapy including cyclosporine, methotrexate, or psoralen with ultraviolet A light (PUVA) in participants with PS
  5. unsatisfactory response despite a full and adequate course of therapy with a corticosteroid and/or an immunosuppressant; or intolerance or medical contraindications for such therapies in CD
  6. unsatisfactory response to conventional therapy including corticosteroids and 6-mercaptopurine (6-MP) or azathioprine (AZA), or intolerance to or medical contraindications for such therapies in UC

Exclusion Criteria:

* Participants who are not covered in the latest version of the adalimumab Summary of Product Characteristics (SPC) for the syringe and pen
* Participants currently enrolled in another study program or clinical trial
* Participants who have been treated with adalimumab before

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants currently being managed in a specialist rheumatology practice or respective hospital department
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-02-05; Primary Completion 2017-08-13 (Actual); Study Completion 2017-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander P Dorr, PhD, Study Director — AbbVie Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants
Period: Overall Study
Arm/Group | Participants Receiving Adalimumab
Started | 96
Completed | 74
Not Completed | 22
Not completed — Lost to Follow-up | 9
Not completed — Lack of Efficacy | 8
Not completed — Serious Adverse Event | 1
Not completed — Participant moved to Germany | 1
Not completed — Aggravation of NY Heart Assoc 3 status | 1
Not completed — Exanthema | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.99 (14.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 96
  More than one race | 0
  Unknown or Not Reported | 0
Number of participants per disease subgroup [Count of Participants; unit: Participants]
  Rheumatoid arthritis (RA) | 42
  Ankylosing spondylitis (AS) | 29
  Plaque psoriasis (PS) | 13
  Psoriatic arthritis (PsA) | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Beliefs About Medicines Questionnaire (BMQ) Specific Score at 12 Months
Description: The BMQ-Specific Scale comprises two 5-item factors assessing beliefs about the necessity of prescribed medication (Specific-Necessity) and concerns about prescribed medication based on beliefs about the danger of dependence, long-term toxicity, and the disruptive effects of medication (Specific-Concerns). Individual items are scored on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 10 (lowest score) to 50 (highest score). Higher scores indicate stronger beliefs.
Time Frame: Baseline and 12 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 72
units on a scale | -1.4 (5.0)

2. Primary Outcome: Correlation Between Beliefs About Medicines Questionnaire (BMQ) Specific Score and Adherence to Treatment as Measured by the Morisky Medication Adherence Scale (MMAS) at 12 Months
Description: The BMQ-Specific Scale comprises two 5-item factors assessing beliefs about the necessity of prescribed medication (Specific-Necessity) and concerns about prescribed medication based on beliefs about the danger of dependence, long-term toxicity, and the disruptive effects of medication (Specific-Concerns). Individual items are scored on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 10 (lowest score) to 50 (highest score). Higher scores indicate stronger beliefs. The MMAS is a 4-item self-reported measure of medication-taking behavior. It measures intentional and non-intentional non-adherence (based on forgetting, carelessness, stopping medication when feeling better, or stopping medication when feeling worse). The MMAS consists of 4 questions which can be answered with yes (0) and no (1). The MMAS score is the sum of all four questions and ranges from 0 (non-adherent) to 4 (adherent).
Time Frame: Baseline and 12 months
Population: Participants with available data
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 73
Spearman correlation coefficient | -.173

3. Secondary Outcome: Change in Morisky Medication Adherence Scale (MMAS) Scores From Month 3 to Month 12
Description: The MMAS is a 4-item self-reported measure of medication-taking behavior. It measures intentional and non-intentional non-adherence (based on forgetting, carelessness, stopping medication when feeling better, or stopping medication when feeling worse). The MMAS consists of 4 questions which can be answered with yes (0) and no (1). The MMAS score is the sum of all four questions and ranges from 0 (non-adherent) to 4 (adherent).
Time Frame: At Month 3 and Month 12
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 77
units on a scale | 0.2 (0.9)

4. Secondary Outcome: Change in the Treatment Satisfaction Questionnaire for Medication (TSQM) Scores From Month 3 to Month 12
Description: The 11-item Treatment Satisfaction Questionnaire for Medication (TSQM) Version II is an instrument to assess participants' satisfaction with medication, providing scores on four scales (side effects, effectiveness, convenience, and global satisfaction). The 11 questions can be answered either with yes/no or by means of a five or seven stage scale (ranging from very unsatisfied to satisfied). TSQM Scale scores range from 0 to 100 and higher scores represent higher satisfaction.
Time Frame: At Month 3 and Month 12
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 77
units on a scale
  Efficacy: number analyzed (Participants) | 76
  Efficacy | 6.80 (23.52)
  Side Effects | 1.95 (17.72)
  Convenience | 3.46 (16.50)
  Global Satisfaction: number analyzed (Participants) | 66
  Global Satisfaction | 3.28 (24.45)

5. Secondary Outcome: Change in Rheumatoid Arthritis Disease Activity Index (RADAI) Scores Over Time
Description: The RADAI is a questionnaire for participants used for measuring disease activity. The index consists of 6 questions. The items ask the participants about (1) global disease activity in the last 6 months, (2) disease activity in terms of current swollen and tender joints, (3) arthritis pain, (4) the current status of health, (5) duration of morning stiffness, and (6) tender joints rated on a joint list. The joint list asks about pain in the left and right shoulders, elbows, wrists, fingers, hips, knees, ankles and toes. The first 4 items are rated on a numeric rating scale from 0 to 10, where higher scores indicate more disease activity. The scores on the last 2 items range from 0 to 6 and 0 to 48, respectively, but are transformed on the same scale of 0 to 10. The RADAI total score is the sum of individual items divided by 5 (range 0-10), with a higher score signifying more disease activity.
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12
Population: Participants with rheumatoid arthritis with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 53
units on a scale
  Baseline | 5.52 (1.66)
  Month 3: number analyzed (Participants) | 47
  Month 3 | 3.99 (1.64)
  Month 6: number analyzed (Participants) | 37
  Month 6 | 2.75 (1.58)
  Month 9: number analyzed (Participants) | 35
  Month 9 | 1.83 (1.64)
  Month 12: number analyzed (Participants) | 39
  Month 12 | 1.86 (1.79)

6. Secondary Outcome: Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score Over Time
Description: The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) assesses disease activity by asking the participant to answer 6 questions (each on a 10 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12
Population: Participants with ankylosing spondylitis with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 28
units on a scale
  Baseline | 5.39 (1.52)
  Month 3: number analyzed (Participants) | 25
  Month 3 | 3.61 (2.05)
  Month 6: number analyzed (Participants) | 24
  Month 6 | 2.98 (1.96)
  Month 9: number analyzed (Participants) | 20
  Month 9 | 1.72 (1.44)
  Month 12: number analyzed (Participants) | 26
  Month 12 | 2.34 (2.30)

7. Secondary Outcome: Change in C-reactive Protein (CRP) Concentration Over Time
Description: C-reactive protein (CRP) was measured from blood samples as a marker for inflammation. Higher levels are indicative of more inflammation. Normal concentration in healthy individuals is usually lower than 1 mg/dL, slightly increasing with age, and increased in a variety of disorders such as rheumatic diseases.
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 90
mg/dL
  Baseline | 1.60 (2.75)
  Month 3: number analyzed (Participants) | 81
  Month 3 | 0.87 (1.66)
  Month 6: number analyzed (Participants) | 70
  Month 6 | 1.54 (8.68)
  Month 9: number analyzed (Participants) | 66
  Month 9 | 0.47 (0.74)
  Month 12: number analyzed (Participants) | 88
  Month 12 | 0.65 (1.25)

8. Secondary Outcome: Changes in Erythrocyte Sedimentation Rate (ESR) Over Time
Description: Erythrocyte sedimentation rate (ESR) indirectly measures how much inflammation is in the body, and is based on the sedimentation and aggregation of erythrocytes (red blood cells). A higher ESR is indicative of increased inflammation. The normal range in healthy individuals is 0 - 10 mm/h for men and 0-15 mm/h for women.
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 86
mm/hr
  Baseline | 29.3 (23.7)
  Month 3: number analyzed (Participants) | 68
  Month 3 | 24.1 (20.5)
  Month 6: number analyzed (Participants) | 64
  Month 6 | 17.4 (15.8)
  Month 9: number analyzed (Participants) | 61
  Month 9 | 17.8 (18.9)
  Month 12: number analyzed (Participants) | 78
  Month 12 | 16.0 (16.7)

9. Secondary Outcome: Change in Psoriasis Area and Severity Index (PASI) Score Over Time
Description: The Psoriasis Area and Severity Index (PASI) is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12
Population: Participants with psoriasis with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 12
units on a scale
  Baseline | 18.0 (11.5)
  Month 3 | 5.1 (6.6)
  Month 6: number analyzed (Participants) | 9
  Month 6 | 1.5 (1.9)
  Month 9: number analyzed (Participants) | 7
  Month 9 | 1.8 (2.5)
  Month 12: number analyzed (Participants) | 9
  Month 12 | 5.9 (6.8)

ADVERSE EVENTS:
Time Frame: Treatment emergent serious adverse events (TESAEs) were collected from the first dose of study drug until 70 days after the last dose of study drug, up to 62 weeks.
Description: TESAEs were collected whether elicited or spontaneously reported by the participant. Nonserious adverse events were not collected for this study.
Arm/Group | Participants Receiving Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/96
Serious Adverse Events (participants affected / at risk) | 1/96
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Adalimumab (N=96)
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT01768858/Prot_SAP_000.pdf